CLINICAL TRIAL: NCT02372916
Title: Progression of Geographic Atrophy and Intravitreal Injections of Ranibizumab Among Treated for Age-related Macular Degeneration
Brief Title: Geographic Atrophy and Intravitreal Ranibizumab Injections
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: University Health Network, Toronto (Other)
Responsible Party: Sponsor
Other Study IDs: 14-8235
Record Dates: First submitted 2015-02-20; First posted 2015-02-26 (Estimated); Last update posted 2015-02-26 (Estimated); Status verified 2015-02

CONDITIONS: Age-related Macular Degeneration; Geographic Atrophy
MeSH Terms: conditions — Macular Degeneration; Geographic Atrophy | interventions — Ranibizumab

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective

GROUPS / COHORTS (3):
- Dry AMD: Patients with pre-existing GA secondary to AMD NOT requiring intravitreal injections (i.e. Dry AMD)
- Wet AMD and treatment-naive: Patients with pre-existing GA and CNV secondary to AMD requiring intravitreal injections (i.e. Exudative AMD) and are treatment-naïve patients
  Interventions: Drug: Ranibizumab
- Wet AMD with history of intravitreal injections: Patients with pre-existing GA and CNV secondary to AMD requiring intravitreal injections (i.e. Exudative AMD) and have received previous intravitreal injections
  Interventions: Drug: Ranibizumab

INTERVENTIONS:
Drug: Ranibizumab — The medication Ranibizumab is routine standard of care for patients with wet AMD, and this is not an aspect of the study that is considered novel intervention
  Groups: Wet AMD and treatment-naive; Wet AMD with history of intravitreal injections

SUMMARY:
Given the aging population who will be affected by wet AMD and lack of effective GA treatment, it is crucial to assess the safety profile of repeated ranibizumab injections in AMD patients with GA, particularly the possible risk of GA development and enlargement. This potential adverse effect has significant implication in the discussions with patients regarding the risks and benefits of AMD treatment and injection frequency. While monthly injections provide slight improvement of visual acuity at 2 years (Martin et al., 2012), the risk of GA enlargement may offset this benefit in visual acuity.

Previous studies assessed the association between intravitreal ranibizumab injections and de novo GA development in injection-naïve eyes (Martin et al, 2012, Querques et al., 2012., Grunwald et al., 2014), rather than GA enlargement in patients with preexisting GA. To the best of the investigators knowledge, there has been no prospective study assessing the association between intravitreal ranibizumab injections and rate of GA progression in patients with pre-existing GA. There is also no prospective study comparing the morphological features of GA between patients who are receiving intravitreal injections and those who are not, nor the concordance of GA enlargement rate between the 2 eyes among patients receiving and not receiving treatment.

ELIGIBILITY:
Inclusion Criteria:

* Age > 50 years old
* Patients with pre-existing GA secondary to AMD NOT requiring intravitreal injections (i.e. Dry AMD)
* Patients with pre-existing GA and CNV secondary to AMD requiring intravitreal injections (i.e. Exudative AMD) and are treatment-naïve patients
* Patients with pre-existing GA and CNV secondary to AMD requiring intravitreal injections (i.e. Exudative AMD) and have received previous intravitreal injections.
* Able to maintain steady fixation in foveal and parafoveal area for fundus imaging Geographic atrophy (GA), both foveal-sparing and foveal GA. Foveal-sparing GA is defined as no GA within 250μm of the centre (Sunness et al. 1999)
* Area of GA can be imaged in its entirety and is not contiguous with areas of peripapillary atrophy
* Adequate media clarity for quality fundus images

Exclusion Criteria:

* Inability to undergo study procedures (e.g. contraindications to intravitreal injections) or attend follow-up visits CNV attributable to other causes than AMD
* Active intraocular inflammation
* Any other retinopathy, including diabetic retinopathy, retinal venous occlusion, epiretinal membrane

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with both dry and wet-AMD
Sampling Method: Probability Sample
Enrollment: 90 (Estimated)
Dates: Start 2014-11; Primary Completion 2016-11 (Estimated)

PRIMARY OUTCOMES:
Geographic atrophy area progression | Every 6 month for total of 2 years
  To assess the association between rate of geographic atrophy (GA) progression in age-related macular degeneration (AMD) and repeated intravitreal ranibizumab injections

SECONDARY OUTCOMES:
Geographic atrophy morphological characteristics | Every 6 month for total of 2 years
  To determine the difference of GA morphological characteristics between AMD patients receiving intravitreal injections and those who are not
Concordance of GA enlargement rate between the two eyes | Every 6 month for total of 2 years
  To determine the concordance of GA enlargement rate between the two eyes for patients with bilateral GA

CONTACTS AND LOCATIONS:
Locations (1):
- Toronto Western Hospital, Toronto, Ontario, Canada